CLINICAL TRIAL: NCT06493552
Title: A Modular, Open Label, Randomized Phase II/III Trial to Assess Efficacy of Combining sEphB4-HSA (EphrinB2 Inhibitor) With Immunotherapy Regimens in Patients With EphrinB2-High Solid Tumors
Brief Title: Modular Trial of sEphB4-HSA in EphrinB2-High Solid Tumors
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Vasgene Therapeutics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2-001
Record Dates: First submitted 2024-06-25; First posted 2024-07-10 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Muscle-Invasive Bladder Carcinoma; Metastatic Urothelial Carcinoma
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — pembrolizumab; Gemcitabine; Cisplatin; enfortumab vedotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- sEphB4-HSA + Pembrolizumab in MIBC (Experimental): sEphB4-HSA shall be started at a dose of 10mg/kg using actual body weight and administered IV over 60 minutes on days 1 and 8 of each cycle as outlined under section 7.1.3.
  Trial treatment may be administered up to 3 days before or after the scheduled Day 1 of each cycle due to administrative reasons. All trial treatments will be administered on an outpatient basis unless the patient has been admitted for another reason and meets all criteria for further therapy.
  Pembrolizumab dose, schedule, delays, and discontinuation of therapy shall be determined by the treating physician in accordance with product label(s), standard of care and institutional policies.
  Treatment will continue until the prespecified number of cycle of therapy are completed or until progression of disease or unacceptable toxicities where specified by the protocol for specific cohort(s).
  Interventions: Drug: SEphB4-HSA; Drug: Pembrolizumab
- Gemcitabine-Cisplatin (GC) or Pembrolizumab Alone in MIBC (Active Comparator): Dose modification, delays and discontinuation of therapy shall be determined by the treating physician in accordance with product label(s), standard of care and institutional policies.
  Interventions: Drug: Pembrolizumab; Drug: Gemcitabine; Drug: Cisplatin
- sEphB4-HSA + Pembrolizumab in Naive mUC (Experimental): sEphB4-HSA shall be started at a dose of 10mg/kg using actual body weight and administered IV over 60 minutes on days 1 and 8 of each cycle as outlined under section 7.1.3.
  Trial treatment may be administered up to 3 days before or after the scheduled Day 1 of each cycle due to administrative reasons. All trial treatments will be administered on an outpatient basis unless the patient has been admitted for another reason and meets all criteria for further therapy.
  Pembrolizumab dose, schedule, delays, and discontinuation of therapy shall be determined by the treating physician in accordance with product label(s), standard of care and institutional policies.
  Treatment will continue until the prespecified number of cycle of therapy are completed or until progression of disease or unacceptable toxicities where specified by the protocol for specific cohort(s).
  Interventions: Drug: SEphB4-HSA; Drug: Pembrolizumab
- Enfortumab Vedotin (EV) + Pembrolizumab in Naive mUC (Active Comparator): Dose modification, delays and discontinuation of therapy shall be determined by the treating physician in accordance with product label(s), standard of care and institutional policies.
  Interventions: Drug: Pembrolizumab; Drug: Enfortumab vedotin

INTERVENTIONS:
Drug: SEphB4-HSA — A recombinant protein comprised of the soluble form of human receptor EphB4 fused to human serum albumin.
  Other Names: sB4HSA
  Arms: sEphB4-HSA + Pembrolizumab in MIBC; sEphB4-HSA + Pembrolizumab in Naive mUC
Drug: Pembrolizumab — Antibody to human PD-1.
  Other Names: Keytruda
Drug: Gemcitabine — A chemotherapy drug used to treat various types of cancer.
  Other Names: GEM, Gemzar
  Arms: Gemcitabine-Cisplatin (GC) or Pembrolizumab Alone in MIBC
Drug: Cisplatin — A type of chemotherapy drug called an alkylating agent used to treat various types of cancer.
  Other Names: CIS
  Arms: Gemcitabine-Cisplatin (GC) or Pembrolizumab Alone in MIBC
Drug: Enfortumab vedotin — Nectin-4-directed antibody and microtubule inhibitor conjugate.
  Other Names: EV, Padcev
  Arms: Enfortumab Vedotin (EV) + Pembrolizumab in Naive mUC

SUMMARY:
Patients with solid tumors that have high expression levels of EphrinB2 are treated with regimens that include EphrinB2 inhibitor, sEphB4-HSA. The primary objective of this study is to demonstrate additive therapeutic benefit for sEphB4-HSA. The secondary objectives are to determine whether the sEphB4-HSA containing regimen is safe and whether the oncological endpoints of importance in each cohort improve as a result of treatment with sEphB4-HSA containing regimen relative to a predefined threshold or to a control arm in the cohort where available. Treatment continues until progression of disease or unacceptable toxicities arise.

DETAILED DESCRIPTION:
The investigators hypothesize that the inhibition of EphrinB2 overcomes the negative prognostic impact of this biomarker and improves the treatment outcomes. It is further hypothesized that this higher level of activity is attributable to the synergistic immune-stimulatory effect of sEphB4-HSA when combined with pembrolizumab.

Cohort A is designed to treat patients with MIBC whose tumors express EphrinB2. Patients in this cohort will be randomized to receive sEphB4-HSA + Pembrolizumab or Gemcitabine-Cisplatin (GC) regimen per standard of care of 4 cycle. Patients ineligible for cisplatin-based chemotherapy or refusing such chemotherapy will be able to receive pembrolizumab alone for 4 cycles based on PURE-01 data showing comparable response rate to chemotherapy with GC regimen.

Cohort B will study the combination of sEphB4-HSA + Pembrolizumab in previously treated mUC, in EphrinB2-high subgroup, a group that in previous studies demonstrated a 52% response rate. In the multi-institutional retrospective series reported by the study team, the expected response rate for anti-PD-L1/PD-1 antibodies is 12% among tumors with high EphrinB2 expression. This represents more than 4-fold improvement in efficacy of immunotherapy if EphrinB2 is inhibited with a mild toxicity profile for the combination. In contrast, EV + Pembrolizumab while effective, has a significant and at times prohibitive toxicity profile. It is also unclear whether EV + Pembrolizumab can deliver the published results in patients with high EphrinB2 expression. Therefore, Cohort B is designed to explore this question.

Upon study entry, participants in either Cohort will be randomly assigned to either sEphB4-HSA + Pembrolizumab or Standard of Care (Control). Study interventions will be administered according to the protocol and participants will be monitored and assessed for safety and efficacy at designated times throughout the study.

ELIGIBILITY:
Inclusion Criteria:

General Inclusion Criteria for Both Arms

* Willing and able to provide informed consent.
* Men and women 18 years of age, or older.
* Must provide the cell block or a minimum of 15 slides from the diagnostic biopsy or archival tissue.
* Tumor tissue must be submitted for molecular profile through a commercial service such as Tempus, CARIS, Foundation One, etc. This must include a PD-L1 assay.
* Tumor must express EphrinB2 as assessed by USC Norris Core Lab.
* Zubrod performance status of less than or equal to 1.
* Women of childbearing potential must use method(s) of contraception. The individual methods of contraception should be determined in consultation with the treating physician or investigator.
* Women of childbearing potential are eligible if serum pregnancy test obtained during screening is negative. Women are also eligible if one of the following criteria is met:

  * Have undergone a documented hysterectomy and/or bilateral oophorectomy; OR
  * Have medically confirmed ovarian failure; OR
  * Achieved postmenopausal status, defined as follows: cessation of regular menses for at least 12 consecutive months with no alternative pathological or physiological cause; OR
  * A serum follicle stimulating hormone (FSH) level within the laboratory's reference range for postmenopausal women.
* Women must not be breastfeeding.
* Men who are sexually active with women of childbearing potential must agree to use 2 contraceptive methods with a failure rate of less than 1% per year.

  o NOTE: Contraception should be continued using two highly effective methods for a period of 120 days after the last dose of treatment.
* Adequate organ function as defined below using baseline laboratory requirements obtained within 14 days prior to randomization:

  * Measured or calculated creatinine clearance (CrCl) greater than or equal to 30 mL/min using the Cockcroft-Gault formula using actual weight (NOT ideal or adjusted weights).
  * WBC ≥2000/uL
  * Neutrophils ≥1500/uL
  * Platelets ≥100x103/uL
  * Hemoglobin ≥9g/dL
  * AST ≤3 x ULN
  * ALT ≤3 x ULN
  * Bilirubin ≤1.5 x ULN

Module A Inclusion Criteria

* Urothelial carcinoma, variant components and differentiations allowed. Pure small cell not allowed.
* cT2 to cT4a N0M0, by TURBT or imaging.
* No systemic therapy for cancer in the previous 12 months.
* Choice of treatment if randomized to the control arm must be declared prior to randomization. If cisplatin ineligible or refusing, pembrolizumab must be approved by patient's insurance prior to randomization.

Module B inclusion Criteria

* Urothelial carcinoma, variant components and differentiations allowed. Pure small cell not allowed.
* Tumor must be Nectin4 non-amplified- testing performed during pre-screening assessment.
* No systemic therapy for cancer in the previous 12 months.
* Measurable disease as defined by RECIST1.1 criteria

Exclusion Criteria:

* Patients with known symptomatic brain metastases requiring systemic corticosteroids. Patients with previously diagnosed brain metastases are eligible if they have completed their treatment and have recovered from the acute effects of radiation therapy or surgery prior to the start of study medication, have discontinued corticosteroid treatment for these metastases for at least 4 weeks and are neurologically stable. Mild neurological deficit is allowed, if it does not interfere with the ability to judge the safety on the trial.
* History of or active autoimmune disorders (including but not limited to: Crohn's Disease, rheumatoid arthritis, scleroderma, systemic lupus erythematosus, Grave's disease) and other conditions that compromise or impair the immune system.
* Known active bacterial, fungal or viral infection including hepatitis B (HBV), hepatitis C (HCV), known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS) -related illness. Routine testing is not required; however, treating physicians may use their discretion to determine whether testing is necessary.
* Uncontrolled adrenal insufficiency.
* Any known active chronic liver disease.
* Concurrent or active second malignancy requiring systemic therapy is excluded.
* Known medical condition (eg, a condition associated with diarrhea or acute diverticulitis) that, in the investigator's opinion, would increase the risk associated with study participation or study drug administration or interfere with the interpretation of safety results.
* Major surgery less than 6 weeks prior to the first dose of study drug. Minor surgery less than 4 weeks prior to the first dose of study drug. Insertion of vascular access device ≥ 7 days prior to 1st dose of study drug is allowed.
* History of severe hypersensitivity reaction to any monoclonal antibody.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2025-03-15 (Actual); Primary Completion 2029-09 (Estimated); Study Completion 2034-08 (Estimated)

PRIMARY OUTCOMES:
Improved pathological response (pCR) in sEphB4-HSA+Pembro vs. Standard of Care for MIBC | Through study completion, an average of 6 months
  Pathologic complete response (pCR), a binary outcome. pCR is defined as absence of the muscle invasive component of the tumor in the radical cystectomy specimen by pathologic review. CIS (pTis), pT1, and pTa are considered to be pCR. All patients with pCR must have pN0/M0. Patients don't have pCR due to refusal of radical cystectomy, dropout prior to radical cystectomry, or pathologic evaluation results are inconclusive or unknown will be classified as non-responders in the ITT.
Improved Overall Survival (OS) in sEphB4-HSA+Pembro vs. Standard of Care for MIBC | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
  Overall survival (OS) defined as period from randomization to death from any cause. OS will be censored at the last follow-up if patients are known to be alive. OS is a time to event variable of the primary interest.
Improved Radiographic Objective Response Rate (ORR) in sEphB4+Pembro vs. Control in mUC | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
  Using RECIST 1.1 on CT or MR imaging of chest, MR imaging of Chest, Abdomen and Pelvis every 6 weeks for the first 3 months and then every 12 weeks.
Non-inferior Overall Survival (OS) of sEphB4+Pembro vs. Control in mUC | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
  Overall survival (OS) defined as period from randomization to death from any cause. OS will be censored at the last follow-up if patients are known to be alive. OS is a time to event variable of the primary interest.

SECONDARY OUTCOMES:
Improved Disease Free Survival and/or Event Free Survival in sEphB4 vs. control for MIBC arm. | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
  Event free survival (EFS): defined as time from randomization to any of the following events: documented disease progression precluding surgery, progression or recurrence diasease after surgery, or death due to any cause. Progresssion/recurrence will be assessed per RECIST 1.1. Patients who undego surgery with incomplete resection will be considered to have an event. Patients who start any subsequent anti-cancer therapy without a prior reported progression/recurrence will be censored at the last evaluable tumor assessment prior to initiation of the subsequent anticancer therapy. Patients who remain free of abovementioned events will be censored at the last follow-up time.
Improved toxicity of EphB4-HSA + Pembro in MIBC vs. control | From start of study intervention until one week after cessation of study intervention, assessed up to 60 months
  Toxicity, as measured by the CTCAE v5.0, will be evaluated from start of study treatment to 7 days after the end of the study treatment.
Improved Duration of Response and/or Progression Free Survival in sEphB4 vs. control for mUC arm. | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
  Disease free survival is defined as the time from the date of surgery to the earlier of disease recurrence, or death from any cause. Disease recurrence includes muscle-invasive recurrences specifically in the bladder, metastatic disease outside the bladder, or death. Patients alive without documented disease recurrence will be censored at the date of last disease assessment. Measured using RECIST 1.1 on CT or MR imaging of chestMR imaging of Chest, Abdomen and Pelvis every 6 weeks for the first 3 months and then every 12 weeks.
Improved toxicity of sEphB4-HSA + Pembro in mUC vs. control | From start of study intervention until one week after cessation of study intervention, assessed up to 60 months
  Toxicity, as measured by the CTCAE v5.0, will be evaluated from start of study treatment to 7 days after the end of the study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Sarmad Sadeghi, MD, Principal Investigator — University of Southern California
Locations (1):
- Sarcoma Oncology Center, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: No